CLINICAL TRIAL: NCT02302976
Title: GLP-1 Agonism for Blocking Cocaine Euphoria and Self-Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Gustavo Angarita, Assistant Professor of Clinical Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1409014655; 1R21DA040914-01A1 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2014-11-27 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine; Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- acute pre-treatment with exenatide (Experimental): This arm plans to explore the effects of acute pre-treatment with the glucagon like peptide-1 (GLP-1) agonist, exenatide vs. placebo, on the subjective (e.g., euphoric) and behavioral effects (e.g., self-administration) of cocaine in experienced, non-treatment seeking users of the drug. We propose to study 24 subjects in a within-subject (two-day, randomized, placebo-controlled) human laboratory study of self-regulated cocaine administration. We hypothesize that acute treatment with exenatide will reduce cocaine-induced euphoria and self-regulated cocaine administration as compared to placebo
  Interventions: Drug: cocaine hydrochloride; Drug: exenatide
- sub-chronic (5 day) treatment with exenatide (Experimental): This arm plans to explore the effects of sub-chronic (5-day) treatment with exenatide as compared to placebo on the subjective (e.g., euphoric) and behavioral (self-administration) effects of cocaine in experienced, non-treatment seeking users of the drug. Upon completion of arm 1, subjects may opt to be randomized to five days of treatment with either exenatide or placebo, followed by a one-day human laboratory study of self-regulated cocaine administration. We hypothesize that subjects treated with exenatide (up to N=12) will demonstrate decreased self-regulated cocaine administration as compared to subjects treated with placebo (up to N=12).
  Interventions: Drug: cocaine hydrochloride; Drug: exenatide
- acute pre-treatment with placebo (Placebo Comparator): This arm plans to explore the effects of acute pre-treatment with the glucagon like peptide-1 (GLP-1) agonist, exenatide vs. placebo, on the subjective (e.g., euphoric) and behavioral effects (e.g., self-administration) of cocaine in experienced, non-treatment seeking users of the drug. We propose to study 24 subjects in a within-subject (two-day, randomized, placebo-controlled) human laboratory study of self-regulated cocaine administration. We hypothesize that acute treatment with exenatide will reduce cocaine-induced euphoria and self-regulated cocaine administration as compared to placebo
  Interventions: Drug: cocaine hydrochloride; Drug: placebo
- sub-chronic (5 day) treatment with placebo (Placebo Comparator): This arm plans to explore the effects of sub-chronic (5-day) treatment with exenatide as compared to placebo on the subjective (e.g., euphoric) and behavioral (self-administration) effects of cocaine in experienced, non-treatment seeking users of the drug. Upon completion of arm 1, subjects may opt to be randomized to five days of treatment with either exenatide or placebo, followed by a one-day human laboratory study of self-regulated cocaine administration. We hypothesize that subjects treated with exenatide (up to N=12) will demonstrate decreased self-regulated cocaine administration as compared to subjects treated with placebo (up to N=12).
  Interventions: Drug: cocaine hydrochloride; Drug: placebo

INTERVENTIONS:
Drug: cocaine hydrochloride
Drug: exenatide
  Other Names: byetta
  Arms: acute pre-treatment with exenatide; sub-chronic (5 day) treatment with exenatide
Drug: placebo
  Arms: acute pre-treatment with placebo; sub-chronic (5 day) treatment with placebo

SUMMARY:
The investigators plan to explore the effects of acute pre-treatment with the glucagon like peptide-1 (GLP-1) agonist, exenatide versus placebo, on the subjective (e.g., euphoric) and behavioral effects (e.g., self-administration) of cocaine in experienced, non-treatment seeking users of the drug. Additionally, the investigators plan to explore the effects of sub-chronic (5-day) treatment with exenatide as compared to placebo on the subjective (e.g., euphoric) and behavioral (self-administration) effects of cocaine in experienced, non-treatment seeking users of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 50 years,
2. voluntary, written, informed consent,
3. physically healthy by medical history, physical, neurological, ECG, and laboratory examinations,
4. DSM-IV criteria for Cocaine Abuse (305.60) or Cocaine Dependence (304.20)
5. recent street cocaine use in excess of amounts to be administered in the current study,
6. intravenous and/or smoked (crack/ freebase) use,
7. positive urine toxicology screen for cocaine,
8. for females, non-lactating, no longer of child-bearing potential (or agree to practice effective contraception during the study), and a negative serum pregnancy (β-HCG) test.

Exclusion Criteria:

1. Other drug dependence (except nicotine) as determined by urine toxicology or interview
2. < 1 year of cocaine dependence,
3. a primary major DSM-IV psychiatric diagnosis (schizophrenia, bipolar disorder, etc.), unrelated to cocaine,
4. a history of significant medical (cardiovascular) or neurological illness, ie prior myocardial infarction, current active symptoms of cardiovascular disease / angina, evidence of cocaine-related cardiovascular symptoms, prior arrhythmias or need for cardiovascular resuscitation, neurovascular events such as transient ischemic attacks, stroke, and/or seizures Parameters re: elevations in vital signs are now explicitly specified under "Safety features built into our one-day self-administration paradigm).
5. current use of psychotropic and/or potentially psychoactive prescription medication,
6. seeking treatment for drug abuse/dependence (for experimental cocaine component),
7. physical or laboratory (β-HCG) evidence of pregnancy.
8. current use of any medication (prescription or over-the-counter) determined to cause potential drug interactions by the study physicians.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-11; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Mean cocaine inter-infusion interval | 3 hours
  Subjects will complete a 90 minute long "binge" cocaine self administration session (16mg/70kg). Mean inter-infusion intervals (time between cocaine boluses) will then be averaged by adding all intervals within the session and dividing by 90. Intervals during which pump access is withheld (due to increase in vital signs) will be excluded. Data on cocaine self-administration (total number of responses, infusions, and III), subjective effects, and vital signs will be checked for normality prior to analysis using Kolmogorov-Smirnov statistics and normal probability plots. The significance level for all statistical tests will be set at p<.05.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Angarita, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States